CLINICAL TRIAL: NCT00492258
Title: SORCE: A Phase III Randomised Double-Blind Study Comparing Sorafenib With Placebo in Patients With Resected Primary Renal Cell Carcinoma at High or Intermediate Risk of Relapse
Brief Title: Sorafenib in Treating Patients at Risk of Relapse After Undergoing Surgery to Remove Kidney Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: MRC-RE05-SORCE; CDR0000553251 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT ID 2006-006079-19; EU-20734; ISRCTN38934710
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2008-04

CONDITIONS: Kidney Cancer
Keywords: stage II renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer; stage I renal cell cancer; clear cell renal cell carcinoma; papillary renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Sorafenib; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: sorafenib tosylate
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving sorafenib after surgery may kill any tumor cells that remain after surgery. It is not yet known whether sorafenib is more effective than a placebo in treating kidney cancer.

PURPOSE: This randomized phase III trial is studying sorafenib to see how well it works compared with a placebo in treating patients at risk of relapse after undergoing surgery to remove kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare disease-free survival of patients with resected primary renal cell carcinoma at high- or intermediate-risk of relapse treated with a placebo for 3 years vs a placebo for 2 years and sorafenib tosylate for 1 year vs sorafenib tosylate for 3 years.

OUTLINE: This is a randomized, placebo-controlled, double-blind, open-label, multicenter study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive oral placebo twice daily for 3 years in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral sorafenib tosylate twice daily for 1 year and oral placebo twice daily for 2 years in the absence of disease progression or unacceptable toxicity.
* Arm III: Patients receive oral sorafenib tosylate twice daily for 3 years in the absence of disease progression or unacceptable toxicity.

Patients in arms I and II with progressive disease may cross over and receive treatment in arm III.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma (RCC)

  * Clear cell or non-clear cell tumors allowed
  * Intermediate- or high-risk disease (Leibovich score 3 to 11)
* Must have undergone surgery for RCC at least 4 weeks but no more than 3 months prior to study entry

  * No evidence of residual macroscopic disease on post-operative CT scan after resection of RCC

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* WBC > 3,400/mm³
* Platelet count > 99,000/mm³
* Creatinine < 2.5 times upper limit of normal (ULN)
* Liver function tests < 1.5 times ULN
* Serum amylase < 1.5 times ULN
* PT/INR < 1.5 times ULN
* PTT < 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 9 months after completion of study treatment
* No cardiovascular conditions, including any of the following:

  * Cardiac arrhythmias requiring anti-arrhythmic medication

    * Beta-blockers and digoxin allowed
  * Symptomatic coronary artery disease or ischemia
  * Myocardial infarction within the past 6 months
  * NYHA class II-IV congestive heart failure
* No active clinically serious bacterial or fungal infection
* No known history of HIV infection
* No chronic hepatitis B or C
* No other prior malignancy except carcinoma in situ of the cervix or adequately treated basal cell carcinoma
* No uncontrolled hypertension

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior treatment for RCC other than nephrectomy
* More than 30 days since prior and no other concurrent investigational therapy
* No concurrent medications that have adverse interactions with sorafenib tosylate including, but not limited to, any of the following:

  * Rifampin
  * Grapefruit juice
  * Ritonavir
  * Ketoconazole
  * Itraconazole
  * Hypericum perforatum (St John's wort)
* No concurrent bone marrow transplant or stem cell rescue
* No other concurrent drug that targets angiogenesis, especially VEGF or VEGF receptors (e.g., bevacizumab)
* No other concurrent drug that targets Ras-pathway or EGFR
* No other concurrent anticancer therapy (chemotherapy, immunotherapy, signal transduction inhibition, or hormonal therapy)
* Concurrent non-conventional therapies (e.g., herbs or acupuncture) and vitamin or mineral supplements allowed
* Concurrent bisphosphonates for prophylaxis of osteoporosis allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1656 (Estimated)
Dates: Start 2007-06; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Disease-free survival

SECONDARY OUTCOMES:
Metastasis-free survival
Disease-specific survival time
Overall survival
Cost effectiveness
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Eisen, Principal Investigator — Cancer Research UK
Locations (39):
- United Kingdom (39):
  - Royal Bournemouth Hospital, Bournemouth, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Queen's Hospital, Burton-on-Trent, England
  - Addenbrooke's Hospital, Cambridge, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Derbyshire Royal Infirmary, Derby, England
  - Dorset County Hospital, Dorchester, England
  - Gloucestershire Royal Hospital, Gloucester, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - Ipswich Hospital, Ipswich, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Lincoln County Hospital, Lincoln, England
  - Saint Bartholomew's Hospital, London, England
  - Medical Research Council Clinical Trials Unit, London, England
  - Guy's Hospital, London, England
  - Royal Marsden - London, London, England
  - Charing Cross Hospital, London, England
  - Maidstone Hospital, Maidstone, England
  - Christie Hospital, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Derriford Hospital, Plymouth, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth Hants, England
  - Whiston Hospital, Prescot Merseyside, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Scarborough General Hospital, Scarborough, England
  - Scunthorpe General Hospital, Scunthorpe, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - Southampton General Hospital, Southampton, England
  - University Hospital of North Staffordshire, Stoke-on-Trent, England
  - Torbay Hospital, Torquay, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales

REFERENCES:
- [Derived] Eisen T, Frangou E, Oza B, Ritchie AWS, Smith B, Kaplan R, Davis ID, Stockler MR, Albiges L, Escudier B, Larkin J, Bex A, Joniau S, Hancock B, Hermann GG, Bellmunt J, Hodgkinson E, Stewart GD, Barber J, Brown J, McMenemin R, Nathan P, Pickering LM, Parmar MKB, Meade A. Adjuvant Sorafenib for Renal Cell Carcinoma at Intermediate or High Risk of Relapse: Results From the SORCE Randomized Phase III Intergroup Trial. J Clin Oncol. 2020 Dec 1;38(34):4064-4075. doi: 10.1200/JCO.20.01800. Epub 2020 Oct 14. PMID 33052759
- [Derived] Blinman PL, Davis ID, Martin A, Troon S, Sengupta S, Hovey E, Coskinas X, Kaplan R, Ritchie A, Meade A, Eisen T, Stockler MR. Patients' preferences for adjuvant sorafenib after resection of renal cell carcinoma in the SORCE trial: what makes it worthwhile? Ann Oncol. 2018 Feb 1;29(2):370-376. doi: 10.1093/annonc/mdx715. PMID 29177440
- [Derived] Fairfax BP, Pratap S, Roberts IS, Collier J, Kaplan R, Meade AM, Ritchie AW, Eisen T, Macaulay VM, Protheroe A. Fatal case of sorafenib-associated idiosyncratic hepatotoxicity in the adjuvant treatment of a patient with renal cell carcinoma. BMC Cancer. 2012 Dec 11;12:590. doi: 10.1186/1471-2407-12-590. PMID 23231599